CLINICAL TRIAL: NCT03997045
Title: Effect of Physical Exercise Program During Pregnancy on Urinary Incontinence
Brief Title: Exercise During Pregnancy and Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Marina Vargas Terrones, PhD, Universidad Politecnica de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AFIPE-001
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Pregnancy; Healthy
Keywords: Pregnancy; Physical exercise; Urinary incontinence
MeSH Terms: conditions — Motor Activity; Urinary Incontinence

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Pregnant women receiving usual care and participating in supervised physical exercise program.
  Interventions: Behavioral: Supervised physical exercise program
- Control group (No Intervention): Pregnant women that are receiving usual care but are not participating in supervised physical exercise program.

INTERVENTIONS:
Behavioral: Supervised physical exercise program — Supervised physical conditioning program of two 60-minutes sessions per week during pregnancy, developed from gestational week 20 to 38. Each session consists of 25-30 minutes of cardiovascular exercise,15 minutes of strengthening exercises, 5 minutes of coordination and balance exercises and 10 minutes of pelvic floor muscles training.
  Arms: Intervention group

SUMMARY:
The aim of this study is to examine the effect of a supervised physical exercise program during pregnancy on urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence | Gestational week 36-38
  Urinary incontinence was measured by the International Consultation on Incontinence Questionnaire Short-Form (ICIQ-SF).

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Barakat Carballo, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Research team website — http://afipe.es/embarazo-y-ejercicio.html